CLINICAL TRIAL: NCT03147833
Title: Ingestion of Protein Before Each Night Sleep to Improve Recovery and Performance in Runners
Brief Title: Protein Before Night Sleep to Improve Recovery and Performance in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Hansen, Associate Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1107229216
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sport beverages Protein (Experimental): Intervention group ingesting PROTEIN
  Interventions: Dietary Supplement: Sport beverages Protein
- Sports beverage Carbohydrate (Active Comparator): Placebo group ingesting carbohydrate
  Interventions: Dietary Supplement: Sport beverages Carbohydrate

INTERVENTIONS:
Dietary Supplement: Sport beverages Protein — Beverage ingested before each night sleep during the intervention
  Arms: Sport beverages Protein
Dietary Supplement: Sport beverages Carbohydrate — Beverage ingested before each night sleep during the intervention
  Arms: Sports beverage Carbohydrate

SUMMARY:
32 runners will be randomized into two groups. The duration of the intervention is one week including a strenuous endurance training program. Group 1 receive a protein beverage before each night sleep and Group 2 receive an isocaloric carbohydrate beverage. Performance test before and after the intervention and blood sampling before and during the intervention to check for markers for muscle damage.

ELIGIBILITY:
Inclusion Criteria: VO2max >55 ml O2/kg/min -

Exclusion Criteria:women, smokers

-

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Performance | 8 days
  5 km time trial

SECONDARY OUTCOMES:
Muscle damage | 8 days
  creatine kinase

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided